CLINICAL TRIAL: NCT00418093
Title: A Phase II Evaluation of Oxaliplatin, Gemcitabine and Bevacizumab in Women With Recurrent Mullerian Carcinoma
Brief Title: Oxaliplatin, Gemcitabine and Bevacizumab in Women With Recurrent Mullerian Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: THe study was terminated early due to a lack of accural
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); Eli Lilly and Company (Industry); Sanofi-Synthelabo (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Neil S. Horowitz, MD, Gynecologic Oncologist, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-356
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: mullerian carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Gemcitabine; Oxaliplatin; Bevacizumab

ARMS (1):
- Chemotherapy (Experimental): All patients received oxaliplatin, gemcitabine, and bevacizumab
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine — Given intravenously over 30 minutes on day 1 and day 15 of a 28-day cycle. Participants can continue study treatment as long as there is no disease progression.
Drug: Oxaliplatin — Given intravenously over 2 hours on day 1 and day 15 of a 28-day cycle. Participants can continue study treatment as long as there is no disease progression.
Drug: Bevacizumab — Given intravenously over 30-90 minutes on day 1 and day 15 of a 28-day cycle. Participants can continue study treatment as long as there is no disease progression.

SUMMARY:
The main purpose of this study is to begin to collect information and try to learn whether or not the combination of oxaliplatin, gemcitabine and bevacizumab works in treating women with recurrent mullerian carcinoma. We will also collect more information about the safety and side effects of this combination of drugs. Gemcitabine and oxaliplatin are chemotherapy drugs that kill cancer cells. Bevacizumab is a new anti-cancer drug that works to slow or stop cell growth in cancerous tumors by decreasing the blood supply to the tumors.

DETAILED DESCRIPTION:
* The study treatment is divided into periods called cycles. Each cycle is 28 days long. Participants will be given the study drugs intravenously on day 1 and day 15 of each cycle.
* Gemcitabine will be given first, over a period of 30 minutes. Then oxaliplatin over a period of 2 hours. Finally, bevacizumab will be given over a period of 30 to 90 minutes. Participants will continue study treatment as long as their tumor is not growing and they are not experiencing unacceptable side effects. If the tumor goes away completely, the participant will have 2 more cycle of study treatment.
* Blood will be drawn for routine testing every week during study treatment to check for side effects. Before day 1 and 15 of each cycle the following tests and procedures will be performed: a medical history; complete physical exam; vital signs; blood tests; and urine tests. Before day 1 of every other cycle, the following additional procedures will be performed: A CT scan, x-ray or ultrasound of your abdomen and pelvis; an x-ray of the chest (if required by the study doctor); blood tests; and urine samples.
* If the participant's tumor goes away, they will be asked to return to the clinic for follow-up visits every 3 months for 2 years, then every 6 months for 3 years. At each follow-up visit the following tests and procedures will be performed: medical history; complete physical examination; CT scan, x-ray or ultrasound of the abdomen and pelvis; x-ray of the chest; and other tests if the doctor feels they are needed.
* There is an optional sub-study that six subjects will be asked to take a part in that will give the study doctors important information about the way the body uses and breaks down the study drugs. This sub-study will involve special surgical procedures and scans that will be done during cycle 1 of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent ovarian, fallopian tube, or primary peritoneal carcinoma. Histologic or cytologic confirmation of the original primary tumor is required.
* Must have measurable disease which is defined as at least one lesion that can be accurately measured in at least one dimension. Each lesion must be >20mm when measured by conventional techniques.
* Must have at least one "target lesion" to be used to assess response.
* Platinum-sensitive tumors, defined as a platinum free interval of at least 6 months, and may have had up to two prior treatment regimens.
* Eastern Cooperative Oncology Group score of 0 or 1
* Life expectancy of 12 weeks or longer
* 18 years of age or older
* Adequate bone marrow, renal, neurologic and liver function
* Normal blood coagulation parameters

Exclusion Criteria:

* Chemotherapy within last 3 weeks
* Current, recent (within 4 weeks), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study.
* Known bleeding disorder or coagulopathy, or history of stroke.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study entry or the anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures within 14 days of study entry.
* Significant cardiovascular disease, New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, a history of deep vein thrombosis, or Grade II or greater, clinically significant peripheral vascular disease within 1 year of study entry.
* Urine protein:creatinine ration greater than or equal to 1.0
* History or clinical evidence of central nervous system disease
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who have evidence of disease within last three years.
* More than 2 prior lines of chemotherapy
* Previous treatment with a VEGF targeted inhibitor or antibody
* Serious non-healing wound, ulcer or bone fracture
* Prior radiation therapy to more than one-third of hematopoietic sites.
* History of abdominal fistulas, gastrointestinal perforation, intra-abdominal abscess, or partial bowel obstruction within 6 months
* Pregnant or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-09; Primary Completion 2011-01 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Horowitz, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy Group: Oxaliplatin plus Gemcitabine plus Bevacizumab
Period: Overall Study
Arm/Group | Chemotherapy Group
Started | 19
Completed Study | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Partial Response Rate
Description: Precentage of women who responded to the treatment regimen Response was determined by RECIST criteria
Time Frame: Outcome was assessed every 2 cycles (every 8 weeks) for the duration on study, an average of 4.5 cycles (18 weeks)
Measure: Number; unit: percentage of patients on study
Groups:
- Chemotherapy Group: Oxaliplatin, Gemcitabine, Bevacizumab
Arm/Group | Chemotherapy Group
Number analyzed (Participants) | 19
percentage of patients on study | 68.4
Statistical Analysis 1: Comparison: Chemotherapy Group; Test type: Superiority or Other; Estimation of PR based on Binomial Model — Exact 95% CI for the partial response rate (13/19 = 0.684): 43.4% ~ 87.4%; We did not perform a test. Point estimate of PR and its exact 95% CI based on Binomial Model is provided. Thus there is no p-value to report; Proportion = 0.684, 95% CI 2-sided [0.43 to 0.87] — Point estimate of PR and its exact 95% CI based on Binomial Model
Statistical Analysis 2: Comparison: Chemotherapy Group; Test type: Superiority or Other; Fisher Exact — We did not perform hypothesis test. We made an estimation for a single proportion (partial response) with its two-sided 95% exact Binomial confidence interval; Single Proportion = 0.684, 95% CI 2-sided [0.434 to 0.874] — Estimation of a single proportion (partial response rate) with exact 95% Binomial confidence interval

2. Secondary Outcome: Progression Free Survival
Description: Time participant remains free of progression of her disease. Evaluated by RECIST criteria
Time Frame: Assessed every 2 cycles (every 8 weeks) of chemotherapy until progression of disease is documented with a median duration of follow up of 24 months
Population: 19
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Chemotherapy Group
Number analyzed (Participants) | 19
weeks | 36.9 [12 to 48]

3. Secondary Outcome: Overall Survival
Description: Duration of time participants are alive after enrolling on the study. Assessed by clinical records
Time Frame: Assessed every 3 months until death from disease, other causes, or loss to follow up at a median follow up of 24 months
Population: All patients enrolled
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Chemotherapy Group
Number analyzed (Participants) | 19
weeks | 112.3 [90.4 to 136]

4. Secondary Outcome: Determine the Nature and Degree of Toxicities Following Treatment With Oxaliplatin, Gemcitabine, and Bevacizumab in This Patient Population.
Description: The nature and toxicities of treatment were graded per the National Cancer Institute Common Terminology Criteria of Adverse Events version 3.0 Patients with grade 2 or higher toxicity were reported
Time Frame: Toxicities were assessed every cycle and for up to 30 days after being removed from the trial
Population: All patients enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy Group
Number analyzed (Participants) | 19
percentage of participants | 94.7

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=19)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=19)
Neutropenia (Blood and lymphatic system disorders) | 6 (6)
Fatigue (General disorders) | 7 (7)
Neuropathy (Nervous system disorders) | 5 (5)
Nausea/Vomiting (Gastrointestinal disorders) | 5 (5)
Hypertension (Cardiac disorders) | 2 (2)
Allergic Reaction to Oxaliplatin (Immune system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was closed after enrolling 19 of the 53 projected patient accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No